CLINICAL TRIAL: NCT00153231
Title: Clinical Evaluation of Morbidity and Efficacy of Posterior IVS (Infracoccygeal Sacropexy), in Comparison to the Standard Sacrospinous Suspension in the Surgical Treatment of Vaginal Vault Prolapse by the Vaginal Route.
Brief Title: Posterior IVS Versus Sacrospinous Suspension in Vaginal Vault Prolapse Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SPIC
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Vaginal Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infracoccygeal sacropexy (Experimental): Intervention: IVS
  Interventions: Device: IVS
- Sacrospinofixation (Active Comparator): Intervention: Sacrospinofixation
  Interventions: Procedure: Sacrospinofixation

INTERVENTIONS:
Device: IVS — Infracoccygeal sacropexy
  Arms: Infracoccygeal sacropexy
Procedure: Sacrospinofixation
  Arms: Sacrospinofixation

SUMMARY:
Hypothesis / aims of study The aim of this multicentre study is to evaluate anatomical and functional results of an innovative posterior tape in vaginal prolapse repair by vaginal route, in comparison to the sacrospinous suspension.

Study design, materials and methods This study involves 5 centres in French Public Hospital. Patients will be randomly allocated to be operated by a sacrospinous suspension or by an posterior IVSTM (Tyco Healthcare, France). Prolapse severity will be evaluated using the POP-Q system. In order to evaluate the patient's quality of life, the validated PFDI and the PFIQ questionnaires will be used preoperatively and during follow-up, as well as a validated questionnaire on sexual problems. The difference on early post-operative pain should be 30% (40% for the sacrospinous suspension and 10% for the posterior IVS). Then the estimated number of patient is 40 in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18
* Vaginal vault prolapse of grade 2 or more (POP-Q system)
* Symptomatic prolapse

Exclusion Criteria:

* Patient unable to read French language
* Cystocele without vaginal vault prolapse
* Vaginal vault prolapse of grade 1
* Associated rectal prolapse
* Rectal inflammatory disease (Crohn, RCH).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2003-03; Primary Completion 2005-12 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Early post-operative pain evaluated by a visual analogic pain the next day after the operation.

SECONDARY OUTCOMES:
- Peri-operative morbidity
- Patient satisfaction
- Quality of life
- Post-operative sexuality
- Anatomical cure rate on vaginal vault support

CONTACTS AND LOCATIONS:
Overall Officials: Renaud de Tayrac, MD, Principal Investigator — Hôpital Carémeau, Nimes, France
Locations (1):
- Hôpital Carémeau, Nîmes, France